CLINICAL TRIAL: NCT00253006
Title: A Quantitative Analysis of Protein- and mRNA-Expression of Nitric Oxide Syntheses and Their Functional Role in Human Urothelium
Brief Title: Analysis of Expression of Nitric Oxide Syntheses and Their Functional Role in Human Urothelium
Status: Terminated | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Zealand University Hospital (Other)
Other Study IDs: UA_H_Ka-05104-m
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-10

CONDITIONS: Interstitial Cystitis; Bladder Diseases; Urinary Incontinence
Keywords: NO; mRNA-expression; pathophysiology; painful bladder syndrome
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Bladder Diseases; Urinary Incontinence | interventions — Proteins

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Tissue examination for protein- and mRNA-expression of NO

SUMMARY:
Painful bladder syndrome (PBS)/interstitial cystitis (IC) may be due to the actions of nitric oxide (NO) in the bladder tissue. NO is a gaseous substance with a very short half-life, synthesized by a group of NO-synthase-enzymes in many tissues.

The goal of this study is to illuminate bladder tissue production of NO in individuals with PBS and healthy individuals, by quantification of NO and NO-enzyme expression by different molecular biological methods.

ELIGIBILITY:
Inclusion Criteria:

* PBS/IC according to International Continence Society (ICS)
* Cystoscopy with bladder distension and deep biopsies within last 5 years
* Cystometry within last 5 years
* Normal urine culture within last month

Inclusion Criteria (for control group):

* Benign non-invasive bladder disease
* No PBS/IC
* Normal urine culture
* No functional bladder disease of known nature (ex. infravesical obstruction)

Exclusion Criteria:

* Age under 18 years
* Inability to understand instructions
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bouchelouche, MD, Study Director — Roskilde County University Hospital at Koege, Dept. of Clinical Biochemistry
Locations (1):
- Copenhagen University Hospital at Herlev, Herlev, Denmark

REFERENCES:
- [Background] Birder LA, Wolf-Johnston A, Buffington CA, Roppolo JR, de Groat WC, Kanai AJ. Altered inducible nitric oxide synthase expression and nitric oxide production in the bladder of cats with feline interstitial cystitis. J Urol. 2005 Feb;173(2):625-9. doi: 10.1097/01.ju.0000145900.22849.1d. PMID 15643277
- [Background] Bouchelouche K, Nordling J. Recent developments in the management of interstitial cystitis. Curr Opin Urol. 2003 Jul;13(4):309-13. doi: 10.1097/00042307-200307000-00007. PMID 12811295
- [Background] Logadottir YR, Ehren I, Fall M, Wiklund NP, Peeker R, Hanno PM. Intravesical nitric oxide production discriminates between classic and nonulcer interstitial cystitis. J Urol. 2004 Mar;171(3):1148-50; discussion 50-1. doi: 10.1097/01.ju.0000110501.96416.40. PMID 14767289